CLINICAL TRIAL: NCT06685224
Title: Parasternal Intercostal Muscle Thickness Versus Ultrasound Assessment of Lung Aeration As a Predictor of Weaning from Mechanical Ventilation; a Prospective Observational Study
Brief Title: Prediction of Weaning Outcome from Mechanical Ventilation Using Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, mahmoud hafez, Mahmoud Tarek Hafez, Tanta University
Other Study IDs: Prediction of Weaning Outcome
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-11

CONDITIONS: Assess the Prediction of Successful SBT and Extubation of Trachea by Bedside Lung Ultrasound in Mechanically Ventilated Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Ultrasound Assessment of the aeration of lung tissue and Parasternal Intercostal Muscle Thickness — Examine the predictive value of lung ultrasound in assessing the success of SBTs and tracheal extubation among patients receiving mechanical ventilation in the intensive care unit (ICU)

SUMMARY:
Examine the predictive value of lung ultrasound in assessing the success of SBTs and tracheal extubation among patients receiving mechanical ventilation in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients will be included in the study when the underlying disease that had required intubation is considered by the attending physician as reversed and after fulfilling the criteria of weaning (alertness, and Adequate gas exchange, normal pH levels, low and stable doses of vasoactive drugs, normal electrolyte levels, and a rapid shallow breathing index (RSBI) of 105 breaths per minute per liter or lower ) rendering the patient eligible to a first SBT.

Exclusion Criteria:

* Exclusion criteria include patients aged < 21yrs , patients with tracheostomy, paraplegia with medullar level above T8, cardiac arrhythmias, severe ICU-acquired neuromyopathy, chronic obstructive pulmonary disease with forced expiratory volume <50% of the theoretical predicted value, patients with planned prophylactic noninvasive ventilation after extubation, and patients who had previously failed a SBT

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tanta University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The aim of this prospective observational study is to evaluate the predictive value of parasternal intercostal muscle thickness vs ultrasound assessment of lung aeration for prediction of weaning outcome from mechanical ventilation | 6 months

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Formenti P, Umbrello M, Dres M, Chiumello D. Ultrasonographic assessment of parasternal intercostal muscles during mechanical ventilation. Ann Intensive Care. 2020 Sep 7;10(1):120. doi: 10.1186/s13613-020-00735-y. PMID 32894372
- [Background] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Background] Berger D, Bloechlinger S, von Haehling S, Doehner W, Takala J, Z'Graggen WJ, Schefold JC. Dysfunction of respiratory muscles in critically ill patients on the intensive care unit. J Cachexia Sarcopenia Muscle. 2016 Sep;7(4):403-12. doi: 10.1002/jcsm.12108. Epub 2016 Mar 9. PMID 27030815
- [Background] Penuelas O, Frutos-Vivar F, Fernandez C, Anzueto A, Epstein SK, Apezteguia C, Gonzalez M, Nin N, Raymondos K, Tomicic V, Desmery P, Arabi Y, Pelosi P, Kuiper M, Jibaja M, Matamis D, Ferguson ND, Esteban A; Ventila Group. Characteristics and outcomes of ventilated patients according to time to liberation from mechanical ventilation. Am J Respir Crit Care Med. 2011 Aug 15;184(4):430-7. doi: 10.1164/rccm.201011-1887OC. PMID 21616997
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624